CLINICAL TRIAL: NCT02229708
Title: Targeting Pregnancy-related Weight Gain to Reduce Disparities in Obesity: a Randomized Controlled Trial
Brief Title: Targeting Pregnancy-related Weight Gain to Reduce Disparities in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22201; R40MC26818 (Other Grant/Funding Number: US Department of Health and Human Services, HRSA)
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Pregnancy; Body Weight Changes; Behavioral; Obesity
Keywords: Pregnancy; Weight control; Behavioral; technology-based intervention
MeSH Terms: conditions — Body Weight Changes; Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The Usual Obstetric Care group will receive usual advice about nutrition and activity during pregnancy from their obstetrician along with some additional information about pregnancy and childbirth through readings from The American College of Obstetricians and Gynecologists. In addition, participants will receive weekly text messages to maintain contact and ensure follow-up.
- Healthy Lifestlye Group (Experimental): The Healthy Lifestyle Group will take part in an individual, technology-based behavioral intervention program which will include specific information about nutrition and physical activity, and strategies for helping them make changes to their diet, physical activity, and weight-related behaviors during pregnancy. Participants will receive information through print materials, text messages, a private Facebook group, and in-person visits and phone calls from a health coach who is part of our research team.
  Interventions: Behavioral: Healthy Lifestyle Group

INTERVENTIONS:
Behavioral: Healthy Lifestyle Group
  Arms: Healthy Lifestlye Group

SUMMARY:
The purpose of this study is to find out whether a technology-base healthy lifestyle program is an acceptable and effective way for African-American mothers to improve their eating and activity during pregnancy, compared to usual obstetric care. The goal of the program is to enhance the health of African-American mothers and their babies.

DETAILED DESCRIPTION:
Black women are in particular need for obesity prevention and treatment. The childbearing period represents a critical life stage of heightened vulnerability for new or persistent obesity, especially among Black women, who retain 2-3 times more weight after pregnancy than White women. Pregnancy weight gain is the strongest identified risk factor for retaining a substantial amount of weight after pregnancy, yet few published interventions have been effective in reducing excessive weight gain in pregnancy, particularly among low-income Black mothers.

The proposed research aims to meets the needs of low-income, Black mothers by developing a novel pregnancy intervention that 1) focuses solely on Black women, 2) incorporates Black mothers' information needs, values, and social context, and 3) uses technology to facilitate participant engagement.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant African-American women at least 18 years of age
* BMI at recruitment between 25.0-44.9 kg/m2
* Singleton pregnancy
* Gestational age of ≤ 20 weeks as determined by last menstrual period
* Plan to carry the pregnancy to term and keep the baby
* Own a cell phone with a text messaging plan
* Member of Facebook social networking site
* Able to participate in physical activity
* Participants must be willing to comply with all study-related procedures

Exclusion Criteria:

* 1. BMI ≤ 24.9 or ≥ 45.0
* Uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure > 95 mmHg). Participants with controlled hypertension on medication for at least three months are allowable.
* Known atherosclerotic cardiovascular disease
* Known congestive heart failure
* Known diabetes mellitus (type 1 or type 2)
* Uncontrolled thyroid disease. Participants with controlled thyroid disease on medication for at least three months are allowable.
* Known cancer
* Any major active rheumatologic, pulmonary, hepatic, dermatologic disease or inflammatory condition requiring steroids or immune modulating medications
* History of testing HIV positive
* Current smoker or tobacco user
* Current or recent history (past 6 months) of drug or alcohol abuse or dependence
* Participation in any weight control or investigational drug study within 6 weeks of screening
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety for successful participation in the study
* Gastrointestinal Disorders (gallbladder disease, Crohn's disease, etc)
* Previous weight loss surgery
* History of bulimia or anorexia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2014-09; Primary Completion 2017-07-16 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change in maternal weight from early pregnancy to 6 months and 1 year postpartum | Approximately 18 months

SECONDARY OUTCOMES:
Change in maternal cardiometabolic risk factors (glucose tolerance, blood pressure) from early pregnancy to 6 months and 1 year postpartum | Approximately 18 months
Change in infant weight and length from birth to 6 months and 1 year of age | Approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon J Herring, MD, MPH, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States